CLINICAL TRIAL: NCT06936826
Title: Development of a Medical Screening Process for Patients With Acute Psychiatric Symptoms Presenting to the Emergency Department - Protocol for a Modified International Delphi Process
Brief Title: Protocol of an International Delphi Process
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01162;am24Nickel
Record Dates: First submitted 2025-04-08; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Delphi Process; Psychiatric Emergency; Medical Screening

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Delphi Consensus Process — Round 1: Evaluation of current Medical Screening Tools and Scoping Review Results Round 2: Rating previous Statements from Round 1 Round 3: Consensus Round 4: Testing Content and Construct Validity of the new Medical Screening Tool with Clinical Vignettes

SUMMARY:
The aim of this study is to develop a consensus-based protocol for medical screening in patients presenting with acute psychiatric symptoms. Using the Delphi method, the study seeks to identify which medical evaluations should be performed routinely in this patient population and under what circumstances. By engaging a panel of experts, the study aims to reduce variability in current practice and support the development of a standardized, evidence-informed approach.

DETAILED DESCRIPTION:
Background

Patients presenting with acute psychiatric symptoms often require urgent assessment and care. While these symptoms are sometimes the result of a primary psychiatric disorder, they can also stem from or be complicated by underlying medical conditions. Timely and accurate medical screening is therefore essential to rule out or address such conditions before initiating or continuing psychiatric treatment.

Currently, there is no universally accepted standard for how and when to perform medical screening in this context. Practices vary widely between institutions, clinicians, and healthcare systems. Some patients may undergo extensive laboratory testing and physical examinations, while others may receive minimal screening. This lack of standardization can lead to both over- and under-investigation, resulting in unnecessary costs, missed diagnoses, or delays in psychiatric care.

Given these challenges, developing a consensus among experts is a necessary step toward ensuring consistent, safe, and effective care. The Delphi method offers a structured, transparent way to gather and refine expert opinion where strong evidence is lacking or practice is inconsistent.

Study Design

The study uses a modified Delphi approach, involving a structured, multi-round survey process with a panel of experts in psychiatry, emergency medicine, and patient representatives. The goal is to develop a consensus on key elements of medical screening for patients with acute psychiatric symptoms. The process includes four rounds:

Round 1: Exploratory Open-Ended Survey Experts are invited to provide free-text responses on which medical evaluations they consider essential in different clinical scenarios. This round is designed to gather a wide range of ideas and perspectives without imposing predefined categories.

Round 2: Structured Rating of Statements Based on the input from Round 1, the research team compiles a set of statements describing specific medical screening procedures or criteria. Experts are then asked to rate their agreement with each statement on a Likert scale. This helps to identify areas of preliminary consensus and disagreement.

Round 3: Re-evaluation and Feedback Statements that did not reach consensus in Round 2 are re-presented, along with anonymous summary statistics and comments from the previous round. Experts are asked to reconsider their ratings in light of this feedback. This round is intended to move the group closer to consensus.

Round 4: Final Prioritization In the final round, the remaining statements are ranked or rated for priority, clarity, and clinical utility. The goal is to finalize a core set of recommendations that reflect expert consensus and are suitable for implementation in clinical practice.

Throughout the process, responses are collected anonymously to minimize bias and ensure that all participants can express their views freely. The results will inform the development of a standardized protocol that can improve medical screening practices and patient outcomes in acute psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

* proficient in English
* possess prior experience with medical screening processes in the Emergency Department

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: interdisciplinary group from national and international societies in emergency medicine and psychiatry on 5 continents and patient representatives
  * Patient representatives: at least 6 in total; can include patients, patient relatives, caregivers, organizations, experts, or advocates
  * society representatives: national and international societies for emergency medicine and psychiatry from North America, South America, Europe, and Australasia, 3 representatives per region, at least 12 in total; strong interest in medical screening with a proven track record in emergency psychiatry and/or current employment in an emergency psychiatry setting
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Consensus regarding items for the new medical screening tool | through study completion, an average of 7 months
  Consensus is define as agreement over a pre-set benchmark of ≥80% agreement. If ≥80% of the responses of all participants to a variable indicate "agree", "strongly agree" or "very strongly agree" in the final round of this Delphi study, it is considered consensus that the variable will be kept.

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Nickel, Prof. MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Unlu L, Carpenter CR, Sterzer P, Griese JA, Chrobok L, Minotti B, Christ M, Nordstrom K, Skinner C, Lunardi C, Alsma J, Bingisser R, Wilson MP, Nickel CH. Development of a medical screening process for patients with acute psychiatric symptoms presenting to the emergency department: protocol for a modified international Delphi study. BMJ Open. 2025 Oct 20;15(10):e105062. doi: 10.1136/bmjopen-2025-105062. PMID 41120177